CLINICAL TRIAL: NCT04472416
Title: Impact of Virtual Reality Distraction on Pain and Anxiety for Bedside Abdominal VAC Dressing Change - A Randomized Controlled Clinical Trial (VIRPA)
Brief Title: Impact of Virtual Reality Distraction on Pain and Anxiety for Bedside Abdominal VAC Dressing Change
Acronym: VIRPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Prof., University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00091
Record Dates: First submitted 2020-06-30; First posted 2020-07-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pain; Anxiety; Satisfaction, Patient
Keywords: Virtual reality; Pain; Anxiety; Satisfaction; VAC dressing change
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Monocentric non-blinded superiority randomized controlled trial: standardized analgesic protocol + virtual reality device vs. standardized analgesic protocol alone for abdominal VAC dressing change.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized analgesic protocol alone (No Intervention): Abdominal VAC dressing change using an standardized analgesic protocol alone.
- VRD + standardized analgesic protocol (Experimental): Abdominal VAC dressing change using standardized analgesic protocol + virtual reality device
  Interventions: Device: VRD in addition to standardized analgesic protocol

INTERVENTIONS:
Device: VRD in addition to standardized analgesic protocol — Use of VRD in addition to standardized analgesic protoco for abdominal VAC dressing change
  Arms: VRD + standardized analgesic protocol

SUMMARY:
We aim to study the use of a virtual reality device (VRD) in addition to our standardized analgesic care protocol for abdominal bedside VAC dressing change and we hypothesize to decrease pain and anxiety and to increase patients' comfort by this intervention.

DETAILED DESCRIPTION:
Monocentric non-blinded superiority randomized controlled trial: standardized analgesic protocol + virtual reality device vs. standardized analgesic protocol alone for abdominal VAC dressing change.

The day of the procedure, each patient will receive a standardized local and systemic analgesia 30 minutes before starting the procedure. The referring surgeon will explain at this moment every step of the procedure of bedside abdominal VAC dressing change.

Baseline levels of pain and anxiety will be assessed by use of VAS (0-10) and one additional questionnaire (STAI).

Virtual reality device will be activated 15 minutes before the beginning of the procedure and will remain as long as the procedure is going on and for 15minutes after finishing the wound dressing.

15 minutes after removing the VRD and 30minutes after finishing the wound dressing the STAI questionnaire and VAS for anxiety, pain and satisfaction (0-10) will be completed by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a bedside abdominal VAC dressing change
* Patients above 18 years old
* Patients able to give informed consent as documented by signature

Exclusion Criteria:

* Patients under 18 years old
* Patients with impaired cognitive status
* Patients with known psychiatric disorders
* Patients unable to follow the procedures of the study due to language problems
* Not consent provided
* Prior inclusion in the same trial (only 1 VAC dressing change per patient can be studied, the first one)
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change of pain using a virtual reality device in addition to a standardized analgesic protocol for bedside abdominal VAC dressing change. Pain will be measured by using a visual analogue scale (VAS) for pain (0-10) in the two groups. | Baseline (pre-procedure) and immediately after the procedure
  Measurement of pain using a visual analogue scale (VAS) for pain with scores range from 0 (no pain) and 10 (worst possible pain), before (baseline: pre-procedure) and immediately after bedside abdominal vacuum assisted closure (VAC) dressing change in the two groups (virtual reality device + standardized analgesic protocol and standardized analgesic protocol alone) in order to demonstrate if a virtual reality device can reduce pain when used in addition to standard care.

SECONDARY OUTCOMES:
Change of anxiety using a virtual reality device along with a standardized analgesic protocol for bedside abdominal VAC dressing change. Anxiety will be measured by using, in the 2 groups, a VAS scale for anxiety along with a STAI questionnaire. | Baseline (pre-procedure) and immediately after the procedure
  Measurement of anxiety using the validated questionnaire State Trait Anxiety Inventory (STAI) and a visual analogue scale (VAS) for anxiety from 0 (no anxiety) and 10 (worst possible anxiety), before (baseline: pre-procedure) and immediately after bedside abdominal vacuum assisted closure (VAC) in dressing change in the two groups (virtual reality device + standardized analgesic protocol and standardized analgesic protocol alone) in order to demonstrate if a virtual reality device can reduce anxiety used in addition to standard care.
Assessment of patients satisfaction using a virtual reality device in addition to a standardized analgesic protocol for bedside abdominal VAC dressing change. Satisfaction will be measured by using a visual analogue scale (VAS) for satisfaction. | Immediately after the procedure
  Satisfaction assessment using a visual analogue scale (VAS) from 1 (not satisfied at all) to 10 (very satisfied) in the two groups (virtual reality device + standardized analgesic protocol and standardized analgesic protocol alone) in order to demonstrate if a virtual reality device can increase patients satisfaction when used in addition to standard care. The assessment will be performed immediately after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hubner, Prof, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Leavitt T, Bayer LR, Orgill DP. Effect of negative pressure wound therapy on wound healing. Curr Probl Surg. 2014 Jul;51(7):301-31. doi: 10.1067/j.cpsurg.2014.04.001. Epub 2014 Apr 26. PMID 24935079
- [Background] Ma Z, Shou K, Li Z, Jian C, Qi B, Yu A. Negative pressure wound therapy promotes vessel destabilization and maturation at various stages of wound healing and thus influences wound prognosis. Exp Ther Med. 2016 Apr;11(4):1307-1317. doi: 10.3892/etm.2016.3083. Epub 2016 Feb 17. PMID 27073441
- [Background] Banwell P, Withey S, Holten I. The use of negative pressure to promote healing. Br J Plast Surg. 1998 Jan;51(1):79. doi: 10.1016/s0007-1226(98)80142-2. No abstract available. PMID 9577325
- [Background] Sahebally SM, McKevitt K, Stephens I, Fitzpatrick F, Deasy J, Burke JP, McNamara D. Negative Pressure Wound Therapy for Closed Laparotomy Incisions in General and Colorectal Surgery: A Systematic Review and Meta-analysis. JAMA Surg. 2018 Nov 1;153(11):e183467. doi: 10.1001/jamasurg.2018.3467. Epub 2018 Nov 21. PMID 30267040
- [Background] Donlon NE, Boland PA, Kelly ME, Schmidt K, Cooke F, Neary PM, Barry KM, Reynolds JV. Prophylactic negative wound therapy in laparotomy wounds (PROPEL trial): randomized controlled trial. Int J Colorectal Dis. 2019 Nov;34(11):2003-2010. doi: 10.1007/s00384-019-03398-9. Epub 2019 Sep 16. PMID 31529194
- [Background] Sharar SR, Carrougher GJ, Nakamura D, Hoffman HG, Blough DK, Patterson DR. Factors influencing the efficacy of virtual reality distraction analgesia during postburn physical therapy: preliminary results from 3 ongoing studies. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S43-9. doi: 10.1016/j.apmr.2007.09.004. PMID 18036981
- [Background] Wiederhold MD, Gao K, Wiederhold BK. Clinical use of virtual reality distraction system to reduce anxiety and pain in dental procedures. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):359-65. doi: 10.1089/cyber.2014.0203. PMID 24892198
- [Background] Atzori B, Hoffman HG, Vagnoli L, Patterson DR, Alhalabi W, Messeri A, Lauro Grotto R. Virtual Reality Analgesia During Venipuncture in Pediatric Patients With Onco-Hematological Diseases. Front Psychol. 2018 Dec 20;9:2508. doi: 10.3389/fpsyg.2018.02508. eCollection 2018. PMID 30618938
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113
- [Background] Riva G, Mantovani F, Capideville CS, Preziosa A, Morganti F, Villani D, Gaggioli A, Botella C, Alcaniz M. Affective interactions using virtual reality: the link between presence and emotions. Cyberpsychol Behav. 2007 Feb;10(1):45-56. doi: 10.1089/cpb.2006.9993. PMID 17305448
- [Background] Anderson AP, Mayer MD, Fellows AM, Cowan DR, Hegel MT, Buckey JC. Relaxation with Immersive Natural Scenes Presented Using Virtual Reality. Aerosp Med Hum Perform. 2017 Jun 1;88(6):520-526. doi: 10.3357/AMHP.4747.2017. PMID 28539139
- [Background] Navarro-Haro MV, Lopez-Del-Hoyo Y, Campos D, Linehan MM, Hoffman HG, Garcia-Palacios A, Modrego-Alarcon M, Borao L, Garcia-Campayo J. Meditation experts try Virtual Reality Mindfulness: A pilot study evaluation of the feasibility and acceptability of Virtual Reality to facilitate mindfulness practice in people attending a Mindfulness conference. PLoS One. 2017 Nov 22;12(11):e0187777. doi: 10.1371/journal.pone.0187777. eCollection 2017. PMID 29166665
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Guo C, Deng H, Yang J. Effect of virtual reality distraction on pain among patients with hand injury undergoing dressing change. J Clin Nurs. 2015 Jan;24(1-2):115-20. doi: 10.1111/jocn.12626. Epub 2014 Jun 4. PMID 24899241
- [Background] Karaman D, Erol F, Yilmaz D, Dikmen Y. Investigation of the effect of the virtual reality application on experimental pain severity in healthy. Rev Assoc Med Bras (1992). 2019 Mar;65(3):446-451. doi: 10.1590/1806-9282.65.3.446. Epub 2019 Apr 11. PMID 30994846
- [Background] Ding J, He Y, Chen L, Zhu B, Cai Q, Chen K, Liu G. Virtual reality distraction decreases pain during daily dressing changes following haemorrhoid surgery. J Int Med Res. 2019 Sep;47(9):4380-4388. doi: 10.1177/0300060519857862. Epub 2019 Jul 25. PMID 31342823
- [Background] Umezawa S, Higurashi T, Uchiyama S, Sakai E, Ohkubo H, Endo H, Nonaka T, Nakajima A. Visual distraction alone for the improvement of colonoscopy-related pain and satisfaction. World J Gastroenterol. 2015 Apr 21;21(15):4707-14. doi: 10.3748/wjg.v21.i15.4707. PMID 25914482